CLINICAL TRIAL: NCT03457311
Title: Clinical Phase Ⅲ Study for Development of Oral Galactose Single Point (OGSP) Solution (G.S.P. Oral Solution®)
Brief Title: Clinical Study for Development of Oral Galactose Single Point (OGSP) Solution (G.S.P. Oral Solution®)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Richever Enterprise Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Oral GSP-001
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Galactose Single Point (GSP), Residual Liver Function
Keywords: GSP, oral galactose single point (OGSP)
MeSH Terms: conditions — Pseudohypoparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OGSP measurement (Other): For the OGSP measurement, subjects will be orally administered with 1.25 ml/kg G.S.P. oral solution (400 mg/ml of galactose). At least 20 ml water will be given to subjects after drinking G.S.P. oral solution within 3 to 5 minutes. Sixty minutes after oral G.S.P. solution, a sample of 0.5 ml of whole blood will be taken from subject's finger for the determination of OGSP value.
  Interventions: Drug: G.S.P. Oral Solution 400 mg/ml

INTERVENTIONS:
Drug: G.S.P. Oral Solution 400 mg/ml — Oral 1.25 ml/kg BW G.S.P. oral solution after fasting for 6 hours.

SUMMARY:
The primary objective is to determine the oral galactose single point (OGSP) cutoff values to discriminate subjects with different hepatic function. The secondary objective is to analyze the correlations between OGSP and other hepatic function assessment methods among this trial subjects.

DETAILED DESCRIPTION:
A novel, simple, clinically useful quantitative liver function test, called the galactose single point (GSP) method, was developed to assess residual liver function by measuring galactose blood concentration 1 hour after galactose was administered (0.5 g/kg). The galactose single point (GSP) method has been used to evaluate liver function in both humans and rats, and GSP concentration has been found to closely reflect changes in enzyme activity and hepatic blood flow. The Federal Drug Administration of the U.S. has recommended the GSP method in its guidelines for industry pharmacokinetics for patients with impaired hepatic function (FDA 2003). The GSP method has also been successfully applied to measure the clearance of drugs that are excreted from the liver but not metabolized, such as promazine and cefoperazone, specifically in patients with various liver diseases. Hu et al. demonstrated that GSP concentration is strongly correlated with the severity of liver disease.

This translate the traditional GSP method to oral galactose single point (OGSP) that will greatly improve the technical simplicity and reduce the burden to patients and will easily applied to patient both in hospital and home to measure the residual liver function.

ELIGIBILITY:
Inclusion Criteria:

Subject must fulfill all of the following criteria to be eligible for the study:

1. Male or female with age between 20-85.
2. Ability and willingness to provide informed consent, adhere to the study visit schedule and complete all study assessments and language specific questionnaires.

Exclusion Criteria:

Any of the following criteria will disqualify the subject from participation:

1. History of serious allergic reaction to galactose and have galactosemia.
2. History of receiving total gastrectomy, subtotal gastrectomy, celiac disease, or small intestinal resection.
3. History of diabetes mellitus.
4. Subjects are children or handicapped people.
5. Subjects with any other reasons considered by the investigator not in the condition to enter into the trial.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-09-09 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Blood concentration of oral galactose | Sixty minutes
  To determine the OGSP cutoff values based on data obtained from this trial to discriminate subjects with different hepatic function